CLINICAL TRIAL: NCT04681521
Title: The Effects of Hot and Cold Compress on Muscle Cramps, Fatigue And Comfort in Hemodialysis Patients: A Placebo Controlled Randomized Trial
Brief Title: Hot and Cold Compress in Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gülşah Kesik, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KA-19143
Record Dates: First submitted 2020-12-15; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Hemodialysis Complication; Muscle Spasm; Fatigue
Keywords: hemodialysis; muscle cramp; fatigue; comfort; nursing care; complementary therapies
MeSH Terms: conditions — Spasm; Fatigue; Muscle Cramp | interventions — Hot Temperature; Methods

STUDY DESIGN:
Intervention Model Description: placebo controlled randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HOT THERAPY:GROUP A (Experimental): Hot Compress Group
  Interventions: Other: Hot and Cold compress, nursing interventions
- COLD THERAPY:GROUP B (Experimental): Cold Compress Group
  Interventions: Other: Hot and Cold compress, nursing interventions
- PLACEBO: GROUP C (Placebo Comparator): Inoperative compress Group
  Interventions: Other: Hot and Cold compress, nursing interventions

INTERVENTIONS:
Other: Hot and Cold compress, nursing interventions — using thermal compress at 38-39 °C (hot) and 15-16 °C (cold) on the distal regions of both lower extremities of the patients

SUMMARY:
Aims and objectives. To examine and compare the effects of hot and cold compresses administration on muscle cramps, fatigue, and comfort in hemodialysis (HD) patients.

Background. Muscle cramps and fatigue are common complications in HD patients and reduce patient comfort. Among the nursing interventions stated for the management of these complications in the literature, hot and cold therapy are remarkable. To the best of our knowledge, the present study is the first research up to date that examined and compared the effects of hot and cold compress administrations on abovementioned complications in HD.

Design. This placebo-controlled randomized trial was conducted in two hemodialysis centers between February and October 2020.

Methods. The study sample consisted of 69 patients, stratified and randomly allocated to two intervention groups and placebo group. For patients of each group, the implementation of the study continued for four weeks, 12 HD sessions.

DETAILED DESCRIPTION:
Hemodialysis (HD) is a common renal replacement therapy used in the treatment of End-Stage Renal Disease (ESRD) worldwide. Although HD is a life-saving treatment for people with ESRD, it causes some acute and chronic complications. Muscle cramps and fatigue are two of the most common complications in HD, and these also cause reducing comfort. Management of complications in HD patients and ensuring an optimal comfort level are pivotal for nurses. According to the literature, recommended nursing practices for the management of cramps in HD patients include hot and cold therapy methods. Besides, preventing cramps can improve comfort by reducing fatigue. Therefore, this study aimed to examine and compare the effects of hot and cold compresses administration on muscle cramps, fatigue, and comfort in hemodialysis (HD) patients.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-65,
* receiving HD treatment for at least six months,
* three days a week with four-hour sessions
* with blood pressure 120/80 mmHg and higher at the beginning of the HD session,
* did not develop intradialytic hypotension in the first two hours of HD,
* hemoglobin value above 8.0 mg/dL,
* having a stable dry weight for the previous month (less than 2 kg change).

Exclusion Criteria:

* receiving intravenous electrolyte replacement during HD session,
* having a condition that prevented hot or cold administration such as diabetic neuropathy, burns, open wounds, and amputation in the lower extremities,
* with an oncological diagnosis or autoimmune disease (rheumatoid arthritis, systemic lupus erythematosus, ankylosing spondylitis, fibromyalgia, etc.),
* refused to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
muscle cramps | 4 weeks
  Throughout the hemodialysis treatment, the patients were monitored in terms of cramp development and cramp development was recorded in the follow-up chart (CEFC). This chart was created by the researcher through literature review. Each involuntary contraction session in the legs of the patients was evaluated as an episode.

SECONDARY OUTCOMES:
Fatigue | 4 weeks
  At the end of each hemodialysis session, the fatigue level of all participants was measured and recorded using the Piper Fatigue Scale.

OTHER OUTCOMES:
Comfort | 4 weeks
  At the end of each hemodialysis session, the comfort level of all participants was measured and recorded using the Hemodialysis Comfort Scale

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Özdemir, Prof. Dr., Study Director — Hacettepe University; Tolga Yıldırım, Assos. Prof., Study Director — Hacettepe University; Cebrail Cebrailov, M.D., Study Chair — Hacettepe University; Gülseren Çeliksöz, M.D., Study Chair — Betamar Dialysis Center
Locations (1):
- Hacettepe University, Ankara, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In the informed consent form presented to the patients at the beginning of the study, it was clearly stated that individual data would be kept confidential. only data based on study results will be shared as scientific content.